CLINICAL TRIAL: NCT06409858
Title: Efficacy Testing of Les Mills Pilates
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Fraser Valley (Other)
Collaborators: Les Mills International (Unknown)
Responsible Party: Principal Investigator, Gillian Hatfield, Associate Professor, University of the Fraser Valley
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 101548
Record Dates: First submitted 2024-05-03; First posted 2024-05-10 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Core Muscle Endurance
MeSH Terms: interventions — Exercise Movement Techniques

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): All participants will receive twice weekly Pilates classes for 8 weeks
  Interventions: Other: Pilates

INTERVENTIONS:
Other: Pilates — Twice-weekly mat Pilates class for 8 weeks, either in person or online (depending on participant availability)

SUMMARY:
Objectives: Determine the effect of an 8-week intervention of the new group fitness program Les Mills Pilates on balance, core stability, abdominal, back, and hip muscle endurance, flexibility, and mood. Research questions: Does doing Les Mills Pilates twice per week for 8 weeks result in: 1) increased balance, 2) increased core stability, 3) increased abdominal, back, and hip muscle endurance, 4) increased flexibility, and 5) improved mood? Intended outcomes: this study will determine the efficacy of a new group fitness program developed by Les Mills International. Results will be used to help refine the program, as well as in marketing of the program.

ELIGIBILITY:
Inclusion Criteria:

* Not participating in regular core training (no more than 10 minutes per session, twice per week)
* Active (150 minutes per week of moderate to vigorous physical activity)

Exclusion Criteria:

* any neurological, cardiovascular, or musculoskeletal conditions that would put them at risk while participating, or be made worse by exercise
* Participants with current lower back pain
* Pregnant participants

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2024-08-16 (Estimated); Study Completion 2024-08-16 (Estimated)

PRIMARY OUTCOMES:
Core endurance (time to failure in seconds) | 8 weeks
  Endurance of the core muscles- abdominals, back extensors, hip extensors, quadriceps- time to hold a plank (abdominals), biering-sorenson test (back extensors), unilateral hip bridge (hip extensors), wall sit (quadriceps) will be recorded. Participants will hold each position until failure. Higher times to reach failure indicate more endurance (better value).

SECONDARY OUTCOMES:
Balance (single leg reach distance in cm) | 8 weeks
  Y-balance test- distance in cm. Higher distances are better outcomes.
Core stability: Sahrmann trunk stability test | 8 weeks
  Sahrmann trunk stability test- maximum level participants can perform with neutral lumbar spine. Level 1 (minimum value) to Level 5 (maximum value). Higher scores are better outcome.
Flexibility in cm | 8 weeks
  Forward reach test. Participants sit with legs extended and reach forward as far as they can. Reach distance is measured. Higher scores are better outcome (more flexibility).
Mood | Daily for 8 weeks
  Perceived motivation, stress and fatigue on 0 (minimum value) -5 (maximum value) Likert scale, where higher numbers indicate more motivation (better outcome), stress (worst outcome), or fatigue (worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Gillian L Hatfield, PhD, Principal Investigator — University of the Fraser Valley

IPD SHARING:
Plan to Share IPD: No